CLINICAL TRIAL: NCT03827512
Title: Assessment of Professional Practices - Arterial Doppler Waveforms Analysis in PAD
Brief Title: Arterial Doppler Waveforms Analysis in PAD
Acronym: APP-Wave-PAD
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Rennes University Hospital (Other)
Collaborators: French Society of Vascular Medicine (Unknown)
Responsible Party: Sponsor
Other Study IDs: 35RC18_30019_APP-Wave-PAD
Record Dates: First submitted 2019-01-30; First posted 2019-02-01 (Actual); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: French Vascular Physicians
Keywords: Vascular physicians; Peripheral artery disease; classification; doppler waveforms; Saint-Bonnet
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Doppler arterial waveforms analysis — terminology used when describing arterial Doppler waveforms

SUMMARY:
The main objective is to evaluate the differences of terminology used when describing arterial doppler waveforms.

To assess the impact of an educational process

DETAILED DESCRIPTION:
Peripheral artery disease (PAD) is a common pathology that affects more than 200 million people worldwide. The prevalence of this pathology is estimated in France at 11% in patients over 40 years old. The Doppler arterial waveforms analysis is an important element to assess the hemodynamic state of a patient and contributes to the diagnosis of the pathology. A number of classifications have been proposed but their use varies from one university to another. We hypothesize that there is a great heterogeneity in the description of the arterial Doppler flow analysis. In addition, a new classification (Saint-Bonnet) has recently been proposed and we will evaluate the effect of the use of this one. The main objective is to evaluate the differences of terminology used when describing arterial Doppler waveforms.

The secondary objectives are: to understand the variations observed and expected (initial, continuous training, place of exercise ...) and to study the effect of a new classification on the heterogeneity of responses.

ELIGIBILITY:
Inclusion Criteria:

* Vascular physicians enrolled in the mailing list of French society of vascular medicine

Exclusion Criteria:

* No exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Vascular physicians enrolled in the mailing list of French society of vascular medicine
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Differences of terminology | through study completion, an average of 1 year
  Number of different terminologies used by the vascular physicians to describe the arterial flows

SECONDARY OUTCOMES:
Effect of a new classification on the heterogeneity of terminology used | through study completion, an average of 1 year
  Comparison of the number of terminology used without classification and the number of terminology used with a classification (Saint-Bonnet)
Variations of description of the arterial Doppler waveforms | through study completion, an average of 1 year
  Significant difference in terms of heterogeneity by region or place of formation

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume MAHE, MD PHD, Principal Investigator — Rennes University Hospital
Locations (1):
- Centre Hospitalier Universitaire de Rennes, Rennes, France